CLINICAL TRIAL: NCT04484584
Title: The Effect of Complex Decongestive Treatment on Edema and Hand Functions in Patients With Distal Radius Fracture
Brief Title: Complex Decongestive Therapy on Distal Radius Fracture
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Altun, MSc,Physotherapist, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: Traumatic Edema
Record Dates: First submitted 2020-07-09; First posted 2020-07-23 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complex Decongestive Therapy Group (CDT): Complex Decongestive Therapy Group: The treatment was applied by a specialist therapist who received CDT training. The study group rehabilitation and CDT application is 1 hour. CDT Treatment Protocol:
  Deep abdominal technique application Neck region CDT application (supraclavicular fossa circular motion-Eflöraj) Circular movements on ipsilateral Axillar lymph nodes Circular movements on bottle neck cubital fossa Front arm bucket pumping pump push MLD application of dorsal and palmar face of the hand to ulnar and radial bundles
  Bandage Treatment (Fingers and hand and forearm bandage): Patients can stay for 6-8 hours or until the next day.
  Patients can do exercises in bandages. The patient is given home education.
  The treatment was made for approximately 30-45 minutes. Patients were given exercise training at home. Orthopedic rehabilitation is the same as the control group.
  Interventions: Other: complex decongestive therapy
- Orthopedic Rehabilitation Group (OR): Orthopedic Rehabilitation Group: The treatment was made for approximately 30-45 minutes. Patients were given exercise training at home.
  Orthopedic Rehabilitation Treatment Protocol:
  Exercises to be done at 4 to 6 weeks: Wrist NEH (at the pain limit),active exercise,Grasp exercise
  Exercises to be done at 6 to 8 weeks: Wrist NEH (at the pain limit),Active assistive / active exercise, Grasp exercise,Supination-pronation exercise. (Opposite baths and classical massage are recommended from orthopedics)
  Exercises to be done at 8 to 10 weeks: Stretching exercises,Finger strengthening spring with Digiflex spring, Power web combo hand finger arm amplifier, Msd theraflex hand exercise dough, Theraband flevbar exercise bar.
  Exercises to be done at 10 to 12 weeks Wrist strengthening exercises, Resistant exercises to all muscles.
  Interventions: Other: complex decongestive therapy

INTERVENTIONS:
Other: complex decongestive therapy — Manual lymphatic drainage Manuel lymphatic drainage therapeutic technique is used for reducing edema and symptoms related with edema by accelerating lymphatic drainage. The aim of massage along the extremity is to provide fluid drainage.Manuel lymphatic drainage stimulates the internal contraction of lymphatic channels. If interstitial space concentration of protein is reduced, it provides drainage of obstructed lymph fluid from local lymph nodes.

SUMMARY:
Trauma results in inflammatory reactions accompanied by high protein edema. Trauma can also reduce the carrying capacity of the lymphatic system below normal lymphatic load, leading to exposure of lymphedema. Cellular wastes accumulated in interstitial fields and prolonged exudation period create a physiological problem. It causes the recovery time of tissues to be completed late and the functional gains to be delayed.

The aim of the study is to investigate the effect of Complex decongestive therapy on traumatic edema, pain and functionality.

DETAILED DESCRIPTION:
Patients are composed of patients who are referred to the physical medicine and rehabilitation clinic. All patients eligible for the study were informed about treatment and possible risks, and a consent form was signed. Determined evaluations were made to the patients. After 3 weeks of treatment, patients will be invited to the controls and the long-term effects of the treatments will be investigated.

Patients with a diameter difference of more than 50 ml between two extremities and patients without Sudeck Atrophy will be included in the treatment.

The study was planned as a single blind with randomized control. The physiotherapist who performed the treatment received manual lymph drainage therapy training.

The patients were distributed to groups with a computer-based data distribution system. While the patients are sent for treatment, they are directed according to the first assessment. The person who performed the assessment and those who received treatment were planned differently.

The primary purpose of the study was to investigate the long-term effectiveness of complex decongestive therapy on traumatic edema, as well as to evaluate long-term hand functions. Other objectives are to investigate the long-term effects on range of motion, muscle strength, grip strength, pain, and daily living activities.

ELIGIBILITY:
Inclusion Criteria:

* Over 45 years
* Unilateral distal radius fracture treated with plaster cast
* Begin treatment after (7-10) days after removing the plaster
* At least 50 mL of the volume difference between the upper extremities
* Having signed the consent form

Exclusion Criteria:

* Associated ulna fracture
* Pathological fracture
* polytrauma
* Bilateral fractures
* With chronic kidney disease
* The presence of infection

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with distal radius fracture
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Volumetric test measurement | at baseline
  Volumetric test measurement is more than 50 mL, edema is considered to be present.
Volumetric test measurement | 4. week
  Volumetric test measurement is more than 50 mL, edema is considered to be present.
Michigan Hand Outcomes Questionnarie | at baseline
  The raw scale score for each of the six scales is the sum of the responses of each scale item. The raw score is converted to a score ranging from 0-100. The MHQ is scored using a general algorithm. The response categories for one of the questions is reversed and re-coded. For the Pain scale, a higher score indicates more pain. For the other five scales, higher scores indicate better hand performance.
Michigan Hand Outcomes Questionnarie | 4. week
  The raw scale score for each of the six scales is the sum of the responses of each scale item. The raw score is converted to a score ranging from 0-100. The MHQ is scored using a general algorithm. The response categories for one of the questions is reversed and re-coded. For the Pain scale, a higher score indicates more pain. For the other five scales, higher scores indicate better hand performance.
Patient Rated Wrist Evaluation | at baseline
  The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of 2 subscales:
  Pain subscale: contains 5 items each of which is further rated from 1-10. The maximum score in this section is 50 and minimum 0 Function subscale: contains total 10 items which are further divided into 2 sections i.e specific activities (having 6 items) and usual activities (having 4 items). The maximum score in this section is 50 and minimum 0.
Patient Rated Wrist Evaluation | 4. week
  The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of 2 subscales:
  Pain subscale: contains 5 items each of which is further rated from 1-10. The maximum score in this section is 50 and minimum 0 Function subscale: contains total 10 items which are further divided into 2 sections i.e specific activities (having 6 items) and usual activities (having 4 items). The maximum score in this section is 50 and minimum 0.
Quick DASH | at baseline
  Quick DASH measures upper extremity functionality. Quick DASH score calculation is made as disability / symptom score: ([n total score / n] -1) x25. The options are 'no difficulty' 'mild difficulty' 'moderate difficulty' severe difficulty 'and' unable '. 'no difficulty' is zero points and 'unable' is four.
Quick DASH | 4. week
  Quick DASH measures upper extremity functionality. Quick DASH score calculation is made as disability / symptom score: ([n total score / n] -1) x25. The options are 'no difficulty' 'mild difficulty' 'moderate difficulty' severe difficulty 'and' unable '. 'no difficulty' is zero points and 'unable' is four.

SECONDARY OUTCOMES:
Myometer test | at baseline
  Myometer test is an electronic device used to measure muscle strength. It is directly proportional to the result of muscle strength. and the result will increase according to the force. 3 evaluations are made and the average is recorded. According to the manufacturer's specifications, the myometer used has a measurement range of 0 to 30kg with an overload rating to 40kg and an accuracy of ± 0.3kg, and is calibrated to within 0.1kg.
Myometer test | 4.week
  Myometer test is an electronic device used to measure muscle strength. It is directly proportional to the result of muscle strength. and the result will increase according to the force. 3 evaluations are made and the average is recorded. According to the manufacturer's specifications, the myometer used has a measurement range of 0 to 30kg with an overload rating to 40kg and an accuracy of ± 0.3kg, and is calibrated to within 0.1kg.
Dynamometer test | at baseline
  A grip strength dynamometer is useful for testing your hand grip strength. for males (in kg): 45-49 < 34.7 34.7-54.5 > 54.5 50-54 < 32.9 32.9-50.7 > 50.7 55-59 < 30.7 30.7-48.5 > 48.5 60-64 < 30.2 30.2-48.0 > 48.0 65-69 < 28.2 28.2-44.0 > 44.0 70-99 < 21.3 21.3-35.1 > 35.1 for females(in kg): 45-49 < 18.6 18.6-32.4 > 32.4 50-54 < 18.1 18.1-31.9 > 31.9 55-59 < 17.7 17.7-31.5 > 31.5 60-64 < 17.2 17.2-31.0 > 31.0 65-69 < 15.4 15.4-27.2 > 27.2 70-99 < 14.7 14.7-24.5 > 24.5
Dynamometer test | 4.week
  A grip strength dynamometer is useful for testing your hand grip strength. for males (in kg): 45-49 < 34.7 34.7-54.5 > 54.5 50-54 < 32.9 32.9-50.7 > 50.7 55-59 < 30.7 30.7-48.5 > 48.5 60-64 < 30.2 30.2-48.0 > 48.0 65-69 < 28.2 28.2-44.0 > 44.0 70-99 < 21.3 21.3-35.1 > 35.1 for females(in kg): 45-49 < 18.6 18.6-32.4 > 32.4 50-54 < 18.1 18.1-31.9 > 31.9 55-59 < 17.7 17.7-31.5 > 31.5 60-64 < 17.2 17.2-31.0 > 31.0 65-69 < 15.4 15.4-27.2 > 27.2 70-99 < 14.7 14.7-24.5 > 24.5

CONTACTS AND LOCATIONS:
Overall Officials: meltem vural, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital; banu aydeniz, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital; tuba Altun, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital; Hasan Kerem Alptekin, Study Director — Bahçeşehir University
Locations (1):
- Bakirkoy Dr. Sadi konuk training and research hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Priganc V, Walter JR, Sublett SH. Edema assessment and management practice patterns among hand therapists: Survey research. J Hand Ther. 2020 Jul-Sep;33(3):378-385. doi: 10.1016/j.jht.2019.04.005. Epub 2019 Oct 14. PMID 31623957
- [Background] Rohner-Spengler M, Frotzler A, Honigmann P, Babst R. Effective Treatment of Posttraumatic and Postoperative Edema in Patients with Ankle and Hindfoot Fractures: A Randomized Controlled Trial Comparing Multilayer Compression Therapy and Intermittent Impulse Compression with the Standard Treatment with Ice. J Bone Joint Surg Am. 2014 Aug 6;96(15):1263-1271. doi: 10.2106/JBJS.K.00939. PMID 25100773
- [Background] Miller LK, Jerosch-Herold C, Shepstone L. Effectiveness of edema management techniques for subacute hand edema: A systematic review. J Hand Ther. 2017 Oct-Dec;30(4):432-446. doi: 10.1016/j.jht.2017.05.011. Epub 2017 Aug 12. PMID 28807598